CLINICAL TRIAL: NCT06812104
Title: A Phase I, Multicenter, Uncontrolled, Open-label, Non-randomized, Dose-escalation Study of KK2845 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Clinical Trial of KK2845 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2845-001
Record Dates: First submitted 2024-12-23; First posted 2025-02-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- KK2845_1 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_1
- KK2845_2 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_2
- KK2845_3 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_3
- KK2845_4 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_4
- KK2845_5 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_5
- KK2845_6 (Experimental): KK2845 will be administered at several dose levels to determine MTD.
  Interventions: Drug: KK2845_6

INTERVENTIONS:
Drug: KK2845_1 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_1
Drug: KK2845_2 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_2
Drug: KK2845_3 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_3
Drug: KK2845_4 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_4
Drug: KK2845_5 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_5
Drug: KK2845_6 — KK2845 will be administered at several dose levels to determine maximum tolerated dose (MTD).
  Arms: KK2845_6

SUMMARY:
This is the first in human study of KK2845. This trial consists of Part 1 (Dose escalation) and Part 2 (Backfill). In Part 1, the maximum tolerated dose (MTD) will be determined while evaluating the safety and tolerability of KK2845 in patients with relapsed or refractory acute myeloid leukemia. Part 2 will collect additional data at tolerated doses of KK2845.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given their free and voluntary written consent to participate in this clinical trial.
2. Patients must be at least 18 years of age at the time consent is obtained.
3. Patients with a confirmed diagnosis of AML according to the WHO classification (2022 edition) by pathological examination at the performing institution conducted as screening test.
4. Patients who meet the following definition of relapsed or refractory. Relapse: Patients with any of the following relapse findings after achieving CR, CRh, or CRi.

   * Myeloblasts >5%
   * Blood blasts reappear in two peripheral blood samples at least one week apart Refractory: Patients who have failed to achieve CR, CRh, or CRi after a sufficient duration of initial intensive chemotherapy or initial treatment with venetoclax or hypomethylating agents.
5. Patients who are considered to have no standard treatment with sustained remission, who have failed to complete a potentially curative treatment, who have no treatment with a promising therapeutic effect, or who have refused standard treatment.
6. Patients with an ECOG PS of 0 to 2 on screening test.
7. Patients with hematopoietic, hepatic, renal, and cardiac function that meet all of the following criteria on screening test.

   * Hematopoietic capacity

     * Neutrophil count greater than 500/mm3 However, even if the neutrophil count is less than 500/mm3, if the principal investigator or sub investigator judges that the neutrophil count is expected to improve, enrollment in this study is acceptable.
   * Liver function

     * AST within 3.0 times the upper reference limit
     * ALT within 3.0 times the upper reference limit
     * T-Bil within 1.5 times the upper limit of the standard
   * Kidney function

     * Creatinine clearance (Cockcroft-gault formula) equal to or greater than 50 mL/min

   However, even if the creatinine clearance calculated using the above formula is less than 50 mL/min, if the value is equal to or greater than 30 mL/min and the serum creatinine level is within 1.5 times the upper limit of the standard value, enrollment in this study is acceptable

   ・Cardiac function
   * LVEF of 50% or more (MUGA or ECHO)
   * QTcF < 450 msec for males and < 480 msec for females
8. Patients who are expected to survive longer than 3 months.
9. Patients who agree to use a method of contraception which is available and effective in their country from (e.g., condom use) from signing informed consent form to 7 months after completion of KK2845 administration in women of child-bearing potential (WOCBP), or from the first KK2845 administration to 4 months after completion of KK2845 administration in male. WOCBP patients must show negativity of serum or urine pregnancy test at screening. Administration should be initiated only after confirmation of negativity of pregnancy test performed before the first administration of KK2845 (Cycle 1 Day 1). However, even in the case of patients with negative pregnancy test, if the possibility of pregnancy cannot be ruled out based on a medical interview, patients cannot enrolled in this study.

Exclusion Criteria:

1. Patients who are diagnosed with APML.
2. Patients suspected extramedullary disease.
3. Patients with a history of malignancy other than those listed in the inclusion criteria or with active malignancy other than those listed in the inclusion criteria (resected localized basal cell carcinoma and localized squamous cell carcinoma of the skin, resected noninvasive cervical cancer, resected noninvasive breast cancer, and cancers for which the last curative treatment was given more than 5 years ago are eligible for enrollment).
4. Patients with white blood cell count greater than 25000/mm3 (If treatment with hydroxyurea results in a white blood cell count of 25000/mm3 or less, enrollment in this study is acceptable) on screening test.
5. Patients who underwent a previous allogeneic hematopoietic stem cell transplant.

   However, enrollment in this trial is permitted if all of the following criteria are met:
   * At least 6 months have elapsed since allogeneic hematopoietic stem cell transplantation as of Cycle 1 Day 1.
   * The patient does not have active acute GvHD of Grade 2 or higher, nor active chronic GvHD of any severity. Acute GvHD is classified according to the MAGIC criteria (Harris et al., 2016), and chronic GvHD is classified according to the NIH criteria (Jagasia et al., 2015), by Grade or severity. Acute GvHD should be graded according to the MAGIC criteria (Harris et al., 2016), and chronic GvHD according to the NIH criteria (Jagasia et al., 2015).
   * At least 4 weeks have elapsed since the donor lymphocyte infusion at Cycle 1 Day 1.
6. Patients who have received anti-tumor therapy such as anticancer agents or radiotherapy (except for patients taking hormone therapy as adjuvant maintenance therapy for breast or prostate cancer prior to the start of study treatment) within the following time periods prior to Cycle 1 Day 1.

   * anticancer agents: 2 weeks (If hydroxyurea is used to control blasts, registration is acceptable for use up to Day -1)
   * Hormone therapy: 2 weeks
   * Radiation therapy: 4 weeks
   * Unapproved medical devices: 4 weeks
7. Patients who received another investigational drug within 4 weeks or 5 times the half-life prior to Cycle 1 Day 1, whichever is shorter.
8. Patients who underwent major surgery (excluding biopsy, central venous catheter insertion, and tooth extractions, etc.) within 4 weeks prior to Cycle 1 Day 1.
9. Patients who received a live vaccine within 4 weeks prior to Cycle 1 Day 1.
10. Patients who have not recovered to Grade 1 or below from an adverse event caused by previously administered anti-tumor therapy.

    However, patients with alopecia or laboratory abnormalities within the range described in the selection criteria or patients experiencing Grade 2 chronic adverse events may be enrolled in this study if the investigator or subinvestigator determines that the safety evaluation of the subject will not be affected.
11. Patients with the following infections.

    * Required systemic treatment (including bacterial, viral, and fungal pathogens)
    * Difficulty for initiating anti-tumor therapy However, patients with infections controlled by antibiotic or antiviral therapy, or patients receiving prophylactic antibiotic or antiviral therapy, may be enrolled in this study.
12. Patients who are suspected SARS-CoV-2 infection (e.g., patients with mild infectious findings and a positive SARS-CoV-2 test without subsequent documentation of a negative test result, patients suspected of ongoing infection based on clinical characteristics).
13. Patients with active interstitial lung disease (including drug-induced pneumonia) or a history of such disease.
14. Patients who have received continuous systemic administration (oral or intravenous) of steroids or other immunosuppressive drugs within 4 weeks prior to Cycle 1 Day 1.

    However, topical, inhalation use, and low-dose corticosteroids (equivalent to 10 mg/day of prednisolone) is acceptable for enrollment in this study.
15. Patients with a history of clinically severe cardiovascular disease (e.g., complete left bundle branch block, uncontrolled ventricular fibrillation, uncontrolled ventricular arrhythmia, angina pectoris, myocardial infarction, prolonged QT syndrome, NYHA grade III or IV congestive heart failure) within 6 months prior to screening test.
16. Patients with a history of arterial thrombosis (e.g., stroke, pulmonary embolism) within 6 months prior to the screening test.
17. Patients with positive for HBV antigen or antibody, HCV antibody, HIV antibody, or HTLV-1 antibody at screening test. However, the following cases are acceptable for enrollment in this clinical trial.

    * HBV test at screening test is negative for HBs antigen and positive for either HBc or HBs antibody or both, but HBV-DNA test is below the lower limit of quantification or below 20 IU/mL (1.3 LogIU/mL).
    * Clear history of hepatitis B vaccination and positive HBs antibody alone.
    * Negative HCV nucleic acid amplification test (HCV-RNA test) with positive HCV antibody test at screening test.
18. Patients with acquired, unclassifiable or hereditary, primary, or secondary immunodeficiency.
19. Patients with a history of Grade 3 or higher allergic reactions to antibody drugs, payloads, or additives to investigational drugs.
20. Patients who are pregnant, lactating (excluded from this study even if lactation is interrupted), potentially pregnant, or wishing to become pregnant during this study period.
21. Patients with psychiatric disorders, central nervous system illnesses (e.g., encephalopathy), or social conditions that are judged to make compliance with the clinical trial difficult or affect obtaining written consent.
22. Other patients who are considered to be undesirable to participate in this study by investigator or subinvestigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Part 1：Dose escalation) | At the end of Cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Number of Adverse Events | Through study completion, an average of 1 year
Blood Drug Concentration | Pre-dose and post-dose at multiple timepoints for each cycle during the intervention (each cycle is 21 days)
Number of ADA (anti-KK2845 antibody) positive Participants | Through study completion, an average of 1 year
Best overall response (CR, CRh, CRi, MLFS, PR, Not evaluable, Relapsed disease, ORR) | Pre-dose for Cycle 1 Day1, Each end of the cycles (each cycle is 21 days), Inspection at Discontinuation
Duration of remission | Through study completion, an average of 1 year
Event-free survival | Through study completion, an average of 1 year
Time to remission | Through study completion, an average of 1 year
Overall Survival | During the treatment and every 12 weeks after study treatment completion (approximately up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Kirin Co., Ltd., Study Director — Kyowa Kirin Co., Ltd.
Locations (10):
- Japan (10):
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyushu University Hospital, Fukuoka
  - Kanazawa University Hospital, Kanazawa
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osaka
  - Saitama Medical University Hospital, Saitama
  - Toranomon Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.